CLINICAL TRIAL: NCT01506154
Title: A Randomized, Multi-Center, Double-Blind, Placebo-Controlled Phase III Trial to Evaluate the Efficacy, Tolerability and Safety of MRX-7EAT Topical Patch in the Treatment of Pain Due to Recent Onset Supraspinatous and/or Subacromial Tendonitis/Bursitis and/or Subdeltoid Bursitis of Shoulder
Brief Title: Safety & Efficacy Study of MRX-7EAT Patch in the Treatment of Pain of the Shoulder
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: MEDRx USA, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MRX-7EAT-2006
Record Dates: First submitted 2012-01-05; First posted 2012-01-09 (Estimated); Last update posted 2018-01-16 (Actual); Status verified 2012-10

CONDITIONS: Bursitis; Tendonitis; Shoulder Pain
Keywords: bursitis/tendonitis and/or subdeltoid bursitis
MeSH Terms: conditions — Bursitis; Tendinopathy; Shoulder Pain

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): Therapy with placebo
  Interventions: Drug: MRX-7EAT
- MRX-7EAT (Experimental): Therapy with experimental drug
  Interventions: Drug: MRX-7EAT

INTERVENTIONS:
Drug: MRX-7EAT — Once daily application of a patch for 14 days

SUMMARY:
A Randomized, Multi-Center, Double-Blind, Placebo-Controlled Phase III Trial to Evaluate the Efficacy, Tolerability and Safety of MRX-7EAT Etodolac-Lidocaine Topical Patch in the Treatment of Pain due to Recent Onset Supraspinatous and/or Subacromial Tendonitis/Bursitis and/or Subdeltoid Bursitis of the Shoulder.

ELIGIBILITY:
Inclusion Criteria:

* Females of child bearing potential must have a negative pregnancy test and be using an adequate method of birth control.
* Subject has a diagnosis of acute supraspinatous or subacromial bursitis/tendonitis and/or subdeltoid bursitis of one shoulder with the onset of the current episode ≥ 24 hours and ≤ 7 days preceding the screening visit.
* Subject has a Current Pain Intensity rated prior to study entry ≥ 6 but ≤ 8 on a Numeric Pain Rating Scale (NPRS).

Exclusion Criteria:

* Subject has a suspected tear in the rotator cuff, calcific tendonitis, adhesive capsulitis, shoulder fractures, bilateral shoulder pain, bilateral tendonitis and/or bursitis of the shoulders, bicipital tendonitis; or orthopedic surgical treatment is required.
* Subject has a positive Drop Arm Test indicative of a suspected tear; a positive O'Brien's Test suggestive of a glenoid labral tear; a positive Apprehension Test which would be indicative of glenohumeral instability; a positive Yergason's Test which would be indicative of bicipital tendonitis.
* Subject had a previous episode of shoulder pain in the same area within two weeks prior to the current episode; history of chronic pain in the target shoulder; history of rotator cuff injury or previous surgery in the same area.
* Subject received passive physical therapy treatments for the pain in the target shoulder within the past 24 hours.
* Subject has used oral pharmacologic treatment less than 5 half-lives before the baseline assessments.
* Subject has used any form of opioid within 24 hours of study entry or use of opioids for 5 or more consecutive days within the 30 days preceding enrollment.
* Subject has received systemic corticosteroids in the 30 days preceding the screening visit; or local injections such as intra-articular, bursal, peritendinous; topical corticosteroids are acceptable unless applied to the target joint; and inhaled or intranasal steroids acceptable (e.g., Flonase®).
* Subject recently initiated sleep medications, muscle relaxants, anticonvulsants or antidepressants (within the past 30 days).
* Subject used TNF alpha blockers or Class 1 anti-arrhythmic drugs within the past 60 days.
* Subject has a history or physical assessment finding of clinically significant GI ulcers or abnormal bleeding, anemia, kidney disease, liver disease, poorly controlled lung, stomach, heart, or other vital organ disease as determined by the study investigator/physician.
* Subject has fibromyalgia, spondyloarthropathies (SpA) or other systemic arthritis such as rheumatoid arthritis. Arthritis typically localized such as gout or osteoarthritis is acceptable as long as it does not affect the injured area.
* Subject has a painful syndrome (e.g. sciatica) or cervical spine disorder leading to a nerve entrapment syndrome or other medical problem that in the investigator's opinion may interfere with pain measurement of the target joint.
* Subject has active skin lesions or disease at the intended site of study medication application, which may be covered by the patch. Skin lesions include open wounds, rash, papules and vesicles; abrasions, lacerations or any break in skin.
* Subject has a history of allergy to etodolac, other NSAIDs, lidocaine or adhesives (e.g., adhesive tape).
* Subject is scheduled for elective surgery or other invasive procedures during the period of study participation.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2011-12; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Mean of all 16 Current Pain Intensity scores collected on Days 4 through 7 on a 0-10 NPRS. | 7 days

CONTACTS AND LOCATIONS:
Overall Officials: Yuji Kuwabara, Study Chair — IL Pharma
Locations (26):
- United States (26):
  - Birmingham, Alabama
  - Scottsdale, Arizona
  - Los Angeles, California
  - San Diego, California
  - Denver, Colorado
  - Clearwater, Florida
  - Coral Gables, Florida
  - Fort Lauderdale, Florida
  - Kissimmee, Florida
  - Lauderdale Lakes, Florida
  - Miami, Florida
  - Orlando, Florida
  - Boise, Idaho
  - Lexington, Kentucky
  - Marrero, Louisiana
  - Southfield, Michigan
  - Raleigh, North Carolina
  - Fargo, North Dakota
  - Zanesville, Ohio
  - Gresham, Oregon
  - Altoona, Pennsylvania
  - Charleston, South Carolina
  - Dallas, Texas
  - El Paso, Texas
  - San Antonio, Texas
  - Temple, Texas